CLINICAL TRIAL: NCT04368663
Title: The Beneficial Effect of the Traditional Japanese Medicine, Keishi-ka-shakuyaku-daio-to（TJ-134）for Patients With Symptomatic Pneumatosis Cystoides
Brief Title: The Beneficial Effect of TJ-134 for Patients With Symptomatic Pneumatosis Cystoides Intestinalis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Chief of Digestive Disease Center, Showa Inan General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ-134
Record Dates: First submitted 2020-04-16; First posted 2020-04-30 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Pneumatosis Cystoides Intestinalis
Keywords: Pneumatosis Cystoides Intestinalis
MeSH Terms: conditions — Pneumatosis Cystoides Intestinalis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TJ-134 group (Active Comparator): The traditional Japanese medicine, Keishi-ka-shakuyaku-daio-to（TJ-134, 7.5g/day), which consists of a mixture of a compound of peony root (6 g), cinnamon bark (4 g), jujube (4 g), glycyrrhiza (2 g), rhubarb (2 g), and ginger (1 g) is administered to enrolled patients for 8 weeks.
  Interventions: Drug: Japanese traditional medicine group
- Lactomin group (Placebo Comparator): Lactomin (3g/day) is administered to enrolled patients for 8 weeks.
  Interventions: Drug: Japanese traditional medicine group

INTERVENTIONS:
Drug: Japanese traditional medicine group — TJ-134 (7.5g/day) or lactomin (3g/day) is administered for 8 weeks.
  Other Names: Lactomin group

SUMMARY:
The traditional Japanese medicine, Keishi-ka-shakuyaku-daio-to is administered to patients with symptomatic pneumatosis cystoides intestinalis (PCI) as compared with lactomin for 8 weeks.

DETAILED DESCRIPTION:
1. Based on endoscopic finding, patients with symptomatic PCI are recruited.
2. After enrollment, abdominal symptoms are evaluated and abdominal CT is performed.
3. Patients were randomized in a 1:1 ratio in blocks of 4 to undergo either the traditional Japanese medicine or lactomin (control). Randomization was carried out by computer-generated random sequences.
4. The traditional Japanese medicine, Keishi-ka-shakuyaku-daio-to（TJ-134, 7.5g/day), which consists of a mixture of a compound of peony root (6 g), cinnamon bark (4 g), jujube (4 g), glycyrrhiza (2 g), rhubarb (2 g), and ginger (1 g) or lactomin (3g/day) is administered to enrolled patients for 8 weeks.
5. After the administration of each drug for 8 weeks, abdominal symptoms are evaluated and abdominal CT is performed again.

ELIGIBILITY:
Inclusion Criteria:

* typical findings of PCI on colonoscopy; Line or pebble like sessile cysts are distributed around the colon with normal overlying mucosa

Exclusion Criteria:

* patients can not take Keishi-ka-shakuyaku-daio-to（TJ-134）

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of computed tomography (CT) findings | at enrollment and 8 weeks after the administration of TJ134
  Change of the intraluminal gas pockets in the colon on CT images before and after the administration of TJ-134

SECONDARY OUTCOMES:
Bloating and abdominal pain | at enrollment and 8 weeks after the administration of TJ134
  Both bloating and abdominal pain are evaluated using visual analogue scale (VAS) score (0-100; 0, none).
Abdominal symptoms | at enrollment and 8 weeks after the administration of TJ134
  Abdominal symptoms were evaluated on the Gastrointestinal Symptoms Rating Scale (GSRS) one a scale of 1 to5 (1 = none).

CONTACTS AND LOCATIONS:
Locations (1):
- Showa Inan General hospital, Komagane, Nagano, Japan

IPD SHARING:
Plan to Share IPD: No